CLINICAL TRIAL: NCT01110551
Title: A Double-Blind Randomized, Placebo-Controlled, Phase I Dose Escalation Study to Investigate the Safety and Immunogenicity of a Tetravalent Chimeric Dengue Vaccine in Healthy Adult Volunteers
Brief Title: Tetravalent Chimeric Dengue Vaccine Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 09-0055; N01AI80003C
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Dengue
Keywords: Dengue, vaccine, flavivirus
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Group 2: low dose ; ID (Experimental): D1: 8 x 10^3, D2: 5 x 10^3, D3: 1 x 10^4, D4: 2 x 10^5 or placebo intradermally on Days 0 and 90.
  Interventions: Drug: Placebo (ID); Biological: Modified Live Tetravalent Chimeric Dengue Vaccine (ID)
- Group 1: low dose; SC (Experimental): D1: 8 x 10^3, D2: 5 x 10^3, D3: 1 x 10^4, D4: 2 x 10^5 or placebo subcutaneously on Days 0 and 90.
  Interventions: Drug: Placebo (SC); Biological: Modified Live Tetravalent Chimeric Dengue Vaccine (SC)
- Group 4: high dose; ID (Experimental): D1: 2 x 10^4, D2: 5 x 10^4, D3: 1 x 10^5, D4: 3 x 10^5 or placebo intradermally on Days 0 and 90.
  Interventions: Drug: Placebo (ID); Biological: Modified Live Tetravalent Chimeric Dengue Vaccine (ID)
- Group 3: high dose; SC (Experimental): D1: 2 x 10^4, D2: 5 x 10^4, D3: 1 x 10^5, D4: 3 x 10^5 or placebo subcutaneously on Days 0 and 90.
  Interventions: Drug: Placebo (SC); Biological: Modified Live Tetravalent Chimeric Dengue Vaccine (SC)

INTERVENTIONS:
Drug: Placebo (SC) — Phosphate buffered saline administered subcutaneously.
  Arms: Group 1: low dose; SC; Group 3: high dose; SC
Drug: Placebo (ID) — Phosphate buffered saline administered intradermally.
  Arms: Group 2: low dose ; ID; Group 4: high dose; ID
Biological: Modified Live Tetravalent Chimeric Dengue Vaccine (SC) — DENVax is a tetravalent dengue vaccine comprised of four recombinant, live attenuated dengue virus strains: DEN-2 PDK-53 (DENVax-2), DEN-2/1 chimera (DENVax-1), DEN-2/3 chimera (DENVax-3) and DEN-2/4 chimera (DENVax-4). The drug product is formulated in buffer and stored frozen. Low dose contains (dose volume 0.1 mL): D1: 8 x 10^3, D2: 5 x 10^3, D3: 1 x 10^4, and D4: 2 x 10^5, total virus dose [plaque forming units (PFU)]: 2.2 x 10^5. High dose contains (dose volume 0.1 mL): D1: 2 x 10^4, D2: 5 x 10^4, D3: 1 x 10^5, and D4: 3 x 10^5, total virus dose (PFU): 4.7 x 10^5. DENVax administered subcutaneously.
  Arms: Group 1: low dose; SC; Group 3: high dose; SC
Biological: Modified Live Tetravalent Chimeric Dengue Vaccine (ID) — DENVax is a tetravalent dengue vaccine comprised of four recombinant, live attenuated dengue virus strains: DEN-2 PDK-53 (DENVax-2), DEN-2/1 chimera (DENVax-1), DEN-2/3 chimera (DENVax-3) and DEN-2/4 chimera (DENVax-4). The drug product is formulated in buffer and stored frozen. Low dose contains (dose volume 0.1 mL): D1: 8 x 10^3, D2: 5 x 10^3, D3: 1 x 10^4, and D4: 2 x 10^5, total virus dose [plaque forming units (PFU)]: 2.2 x 10^5. High dose contains (dose volume 0.1 mL): D1: 2 x 10^4, D2: 5 x 10^4, D3: 1 x 10^5, and D4: 3 x 10^5, total virus dose (PFU): 4.7 x 10^5. DENVax administered intradermally.
  Arms: Group 2: low dose ; ID; Group 4: high dose; ID

SUMMARY:
The purpose of this study is to test the safety and immune response to a live attenuated dengue vaccine that could protect people against all 4 types of dengue virus. Live attenuated means that while this vaccine contains 4 live dengue viruses the viruses have been attenuated (weakened) so as not to cause dengue disease in people. Dengue virus is spread to people by mosquitoes and can cause sickness and even death. Seventy-two subjects between the ages of 18-45 years old will be enrolled in this research study at Saint Louis University Center for Vaccine Development. Participants will be randomly assigned to 1 of 4 groups to receive 2 doses of the study vaccine or placebo (inactive substance). Study procedures include: maintaining a diary to record temperature and side effects, physical exam, electrocardiogram (ECG) (measures the activity of the heart), and blood samples. Participants will be involved in study related procedures for about 10 months.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and immunogenicity of a tetravalent dengue vaccine administered subcutaneously or intradermally. The hypotheses being tested in this study is whether or not a tetravalent dengue vaccine may be safely administered to healthy normal individuals by intradermal (ID) or subcutaneous (SC) injection and provide measurable levels of serum neutralizing antibodies against all four dengue virus serotypes. The study is also designed to compare safety and immunogenicity between routes of administration and dose levels. The primary objective of this study is to evaluate the safety and tolerability of a two-dose regimen tetravalent dengue vaccine administered either SC or ID to healthy adult volunteers. Two dose levels will be tested in a dose-escalation format. Safety and tolerability will be measured by conducting post-vaccination safety assessments including physical examinations, injection site examinations, adverse event monitoring, hematology, blood chemistry, and urine dipstick. The secondary objective of this study is to assess the immunogenicity of the vaccine, in terms of neutralizing antibodies, against all four dengue serotypes when administered at two dose levels by two routes of administration in healthy adults. Titers of serum neutralizing antibodies will be measured at pre-vaccination, after prime and boost vaccinations and assessed by comparing titers at the two dose levels as well as the two routes of administration. In addition, viremia deriving from the attenuated vaccine viruses will be measured on days 0 (baseline), 2, 4, 5/6, 7, 9, 11, and 14 after both prime and boost vaccinations. Levels of neutralizing antibodies will also be measured in samples to be obtained on days 180 and 270 for analysis and submission in a supplement to the study report. This study will enroll 72 healthy flavivirus-negative male and female subjects between the ages of 18 and 45.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 and less than or equal to 45 years old at time of screening.
* In good health as determined by medical history, physical examination including height and weight, and clinical safety laboratory examinations. For creatinine and alkaline phosphatase levels the applicable cut-offs for determination are the upper limits of normal only, as there is no clinical significance associated with results below the lower limits of normal for these laboratory values. For aspartate aminotransferase (AST) and alanine aminotransferase (ALT), the applicable cut-offs for determination are less than 1.5 times the upper limits of normal, as there is no clinical significance associated with results below the lower limits of normal for these laboratory values or with mild elevations above the upper limits of normal.
* Laboratory values not listed in Table 3 which are obtained as part of a reference laboratory pre-determined panel will be considered as acceptable for enrollment if they are either within reference laboratory normal range or within the ranges specified for a grade I AE per the protocol Toxicology Tables in Appendix B. Values within reference laboratory normal ranges or within ranges specified for a grade I AE per the Toxicology Tables in Appendix B will be considered as discussed with the medical monitor and may be enrolled with no further discussion. Values with deviations outside the ranges specified for a grade 1 AE in the Toxciology Tables in Appendix B will be discussed further between the PI and the medical monitor prior to vaccination and assessed for impact on volunteer safety. Urinalyses obtained from female volunteers on their menses may be repeated after their menses have concluded without discussion with the medical monitor. Laboratory values which are not listed in the Toxicology Tables in Appendix B and which are out of the reference laboratory normal range will be discussed with the DMID medical monitor to determine its relevance for safety and impact on enrollment and follow-up vaccinations.
* Blood tests negative for antibodies to human immunodeficiency virus (HIV)-1, Hepatitis C, dengue, West Nile, and negative for Hepatitis B surface antigen.
* No history of dengue or West Nile infection or participation in a previous dengue or West Nile vaccine trial.
* Females of child bearing potential must have a negative urine pregnancy test result during screening and a negative urine pregnancy test immediately prior to vaccination and be willing to use oral, implantable, transdermal or injectable contraceptives or another reliable means of contraception approved by the Investigator (intrauterine device, female condom, diaphragm with spermicidal, cervical cap, use of condom by the sexual partner or a sterile sexual partner, or abstinence) from screening until after the last blood sample (at day 270).
* Willing and able to give written informed consent to participate.
* Willing and able to communicate with the investigator and understand the requirements of the study.
* Electrocardiogram (ECG) in absence of clinical significance (e.g., complete left or right bundle branch block, incomplete left bundle branch block or sustained ventricular arrhythmia, or two premature ventricular contraction's (PVC's) in a row, or ST elevation consistent with ischemia).
* Weight: greater than or equal to 110 lb.
* Access to a fixed or mobile telephone.

Exclusion Criteria:

* Any condition which would limit the subject's ability to complete the study in the opinion of the Investigator.
* Clinically significant hematological, renal, hepatic, pulmonary, central nervous, cardiovascular, thromboembolic, autoimmune, coagulopathic, or gastrointestinal disorders or history of such disorders
* Any history of malignancy with the exception of basal cell carcinoma.
* Previous history , or current diagnosis of diabetes mellitus.
* Pulse >95 or <40 at rest or irregular, systolic blood pressure (bp) >170 or <90 at rest or diastolic bp >90 or <50 at rest, body temperature >100 F, respirations >25 per minute at rest.
* History of allergy to penicillin, neomycin, streptomycin or gentamicin.
* History of hypersensitivity to any vaccine.
* History of previous vaccination with Yellow Fever (YF) vaccine or Japanese Encephalitis (JE) vaccine or planned receipt of either YF or JE vaccine during the course of the study.
* Previous history of infection with dengue or West Nile or seropositive antibody status to dengue or West Nile virus or participation in a vaccine trial for either of these.
* Travel or planned travel to a dengue-endemic area including the Caribbean, Mexico, Central America, South America or Asia during the study period or in the month prior to screening. An updated map of dengue endemic areas is available at the CDC Yellow Book 2010 website (http://wwwnc.cdc.gov/travel/yellowbook/2010/chapter-5/dengue-fever-dengue-hemorrhagic-fever.aspx) and a list of dengue endemic countries is provided in the Manual of Procedures (MOP).
* Travel to a dengue endemic area within 1 month of screening. Volunteers who have a history of recent travel to a dengue endemic area may screen if they have returned to the US 30 or more days prior to the screening visit.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term (at least 2 weeks within the previous 3 months) systemic corticosteroids therapy (at a dose of at least 0.5 mg/kg/day). Intranasal or topical prednisone (or equivalent) are allowed.
* Personal history of recurring migraines or on prescription medication for treatment of recurring headaches or migraines.
* Use of any non-steroidal anti-inflammatory drugs (NSAIDs), including any aspirin-containing products, acetaminophen or systemic, topical, or intranasal antihistamines for the 3 days immediately prior to each vaccination. Systemic antihistamines may not be used at all during the first 21 days after each vaccination.
* During the first 14 days after each vaccination, anti-inflammatory drugs (NSAIDs) or acetaminophen may be used only if the subject has a fever >/= 100 F or if the subject has significant arm pain, myalgia, arthralgia, or headache and only after documenting the symptom in the memory aid. Intranasal or topical antihistamines may be used during the first 14 days after each vaccination only if the subject has significant allergy symptoms such as rhinitis, cough, eye inflammation, or pruritis and only after documenting the symptom in the memory aid. Intranasal or topical antihistamines, NSAIDs or acetaminophen should only be taken after documentation of symptoms or fever in the memory aid and should not be taken prophylactically.
* Receipt of any other investigational product in the month before study entry and during the entire study duration.
* Receipt or planned receipt of any licensed vaccine in the 4 weeks preceding either trial vaccination (2 weeks for inactivated vaccines) or planned receipt of any vaccine in the 4 weeks following each of the trial vaccinations.
* Concurrent or planned participation in any other clinical study during the conduct of this study.
* Receipt of blood products or immunoglobulins 8 weeks before study entry or planned use during the study period.
* Donation of blood 6 weeks before study entry or at any time during the study.
* Laboratory screening test result that is not within protocol specified normal range (Table 3 of protocol).
* Females who are pregnant or lactating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2010-05; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of volunteers overall and in each dose group with unsolicited vaccine-associated adverse events (AEs) in each dose group. | From time the first dose of vaccine is administered until the end of the study (Study Days 0-270 or through termination visit, if terminated early).
Number of volunteers overall and in each dose group with local or systemic vaccine reactogenicity, based on evaluation of solicited adverse events (AEs) recorded on subject memory aids or during clinical assessments. | Through 14 days after prime or boost vaccination.
Number of volunteers overall and in each dose group with vaccine-associated serious adverse events (SAEs). | From time the first dose of vaccine is administered (Day0) until the end of the study (Day 270).

SECONDARY OUTCOMES:
Immunogenicity: geometric mean neutralizing antibody titers (GMT) to each of the 4 dengue serotypes. | At 14, 30, 60, and 90 days after the prime vaccination on Day 0, and at 14 and 30 days after the boost vaccination on Day 90.
Viremia: incidence, duration, and titer of viremia for each of the DENVax vaccine components. | Days 0, 2, 4, 5/6, 7, 9, 11, and 14 after each vaccination.
Immunogenicity: durability of vaccine-induced immune responses based on neutralizing antibody titers to all 4 dengue serotypes. | At 90 days and 180 days after the boost vaccination will be analyzed for inclusion in a supplemental study report.
Immunogenicity: proportion of subjects seroconverting to each of the 4 dengue serotypes, where seroconversion is defined as plaque reduction neutralization assay (PRNT)50 titer greater than or equal to 10. | Days 0 (pre-prime dose), 14, 30, 60, 90 (pre-booster dose), 104 and 120.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University - Center for Vaccine Development, St Louis, Missouri, United States

REFERENCES:
- [Derived] George SL, Wong MA, Dube TJ, Boroughs KL, Stovall JL, Luy BE, Haller AA, Osorio JE, Eggemeyer LM, Irby-Moore S, Frey SE, Huang CY, Stinchcomb DT. Safety and Immunogenicity of a Live Attenuated Tetravalent Dengue Vaccine Candidate in Flavivirus-Naive Adults: A Randomized, Double-Blinded Phase 1 Clinical Trial. J Infect Dis. 2015 Oct 1;212(7):1032-41. doi: 10.1093/infdis/jiv179. Epub 2015 Mar 19. PMID 25791116